CLINICAL TRIAL: NCT00012831
Title: Nurse Managed Clinic for Dementia Patients and Family Caregivers
Status: Completed | Type: Observational
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Collaborators: GRECC (Unknown)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Other Study IDs: NRI 95-143
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2005-12

CONDITIONS: Alzheimer's Disease; Caregivers; Dementia
MeSH Terms: conditions — Alzheimer Disease; Dementia

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1

SUMMARY:
This study evaluates the effectiveness of a nurse-managed interdisciplinary (nursing and occupational therapy) clinic serving community dwelling dementia patients and their spouse caregivers. It is grounded in a nursing self-care model that guides nurses to identify interventions that fit with the capabilities of individual patients and compensate for their specific deficits. The occupational therapy assessment uses the Allen Cognitive Levels that identify the abilities and deficits of a particular functional level so that the strategies and approaches taught to caregivers can be tailored to the specific needs of the patient.

DETAILED DESCRIPTION:
Background:

This study evaluates the effectiveness of a nurse-managed interdisciplinary (nursing and occupational therapy) clinic serving community dwelling dementia patients and their spouse caregivers. It is grounded in a nursing self-care model that guides nurses to identify interventions that fit with the capabilities of individual patients and compensate for their specific deficits. The occupational therapy assessment uses the Allen Cognitive Levels that identify the abilities and deficits of a particular functional level so that the strategies and approaches taught to caregivers can be tailored to the specific needs of the patient.

Objectives:

The ultimate objective of the study is to increase caregiver competence, maintain optimal function of dementia patients, and show that this nurse managed clinical model can improve the quality of life for both the Alzheimer patients and their caregivers in a cost-effective manner.

Methods:

The study is being conducted as a block design, randomized trial of the Dementia Care Clinic (DCC) compared with the standard interdisciplinary GRECC care. A total of 120 dementia patient/spouse caregiver dyads will be enrolled in the study. Twelve dyads are enrolled in each seven-week block during which a clinic visit and four weekly caregiver education sessions are held for each of the two cohort groups. Follow up clinic visits are made at six months and one year. Data collection interviews are conducted before the first clinic visit, and at three, six, and twelve months. Patient depressed mood is measured by the Yesavage Geriatric Depression Scale (GDS). The Revised Memory and Behavior Problems Checklist is used to measure patient behavior changes and the effect of the behaviors on the caregiver. Positive and negative effects of caregiving are measured by the Zarit Burden Interview, the Center of Epidemiological Studies Depression Scale (CES-D), Phillips Beliefs about Caregiving Scale, and brief scales of perceived mastery, preparedness, and competence in caregiving.

The project will employ multiple independent repeated measures analyses of covariance (RMANCOVA) in which pre-intervention levels of the dependent measures under consideration will be controlled as covariates. Group x time interaction effects will also be examined to test for changing effects of the intervention over the study period. Multiple regression analyses will be used to examine the relationship of cost data to subject and experimental factors.

Status:

Recruitment was completed for the study in 2000. Each cohort of patients and their spouse caregivers have been followed for one year. Baseline data is being analyzed and portions have been presented at recent conferences. Study data is currently being analyzed and analysis is scheduled for completion in December of 2001.

ELIGIBILITY:
Inclusion Criteria:

Subjects are veterans with a diagnosis of Alzheimer's Disease, cared for in their homes by spouse caregivers.

Exclusion Criteria:

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Study Completion 2001-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melitta K. Maddox, MSN, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States